CLINICAL TRIAL: NCT07166705
Title: Investigating the Effects of the Metaverse-Based Education Model on Motivation and Academic Achievement in Physiotherapy and Rehabilitation Students: A Randomized Controlled Study
Brief Title: Metaverse-Based Education for Physiotherapy and Rehabilitation Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mesut ERGAN, assistant professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-12-2025/96/7
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Palpation Skills; Physical Therapy Education; Educational Interventions; Health Professions Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metaverse-Based Education Group (Experimental)
  Interventions: Other: Metaverse-Based Education Group
- Distance/Online Education Group (Experimental)
  Interventions: Other: Distance/Online Education Group
- Traditional Face-to-Face Education Group (Experimental)
  Interventions: Other: Traditional Face-to-Face Education Group

INTERVENTIONS:
Other: Metaverse-Based Education Group — As part of this intervention, participants will receive palpation skills training in a metaverse-based virtual learning environment. The training consists of three modules, each of which will cover the palpation of a different anatomical region:
  * Module 1: Cervical region palpation
  * Module 2: Thoracic region palpation
  * Module 3: Lumbo-pelvic region palpation The training will be delivered in a three-dimensional virtual classroom environment using avatars. Participants will engage in interactive exercises based on scenarios structured on the metaverse platform and, under the guidance of an instructor, will practice palpation techniques on virtual patient models.
  Sessions will be conducted in a group format, allowing students to interact with each other in real-time. Voice communication, motion tracking, and virtual feedback mechanisms will be used throughout the training.
  Arms: Metaverse-Based Education Group
Other: Distance/Online Education Group — As part of this intervention, a palpation skills course will be delivered to participants online via the Microsoft Teams application. The training consists of three modules, each of which will cover the palpation of different anatomical regions.
  Module 1: Cervical region palpation Module 2: Thoracic region palpation Module 3: Lumbo-pelvic region palpation The training will utilize theoretical information, visual materials, and live/pre-recorded practice videos. Participants will attend the course as a group and participate in structured learning sessions guided by the instructor in each module.
  Arms: Distance/Online Education Group
Other: Traditional Face-to-Face Education Group — As part of this intervention, participants will be taught palpation skills in a face-to-face classroom setting using traditional teaching methods. The training consists of three modules:
  Module 1: Palpation of the cervical region Module 2: Thoracic region palpation Module 3: Lumbo-pelvic region palpation Throughout the training, the instructor will conduct structured theoretical presentations, demonstrations, and face-to-face practice sessions. Students will observe palpation techniques through live demonstrations by the instructor and then have the opportunity to practice one-on-one.
  Arms: Traditional Face-to-Face Education Group

SUMMARY:
In the modern era, university students, especially those from Generation Z, are true digital natives who have grown up with technology and embraced it wholeheartedly. This hyper-cognitive generation has different characteristics than their predecessors and emphasizes educational approaches integrated with innovative technologies over traditional methods. Rather than traditional classroom learning, Generation Z prefers to learn through various media, such as digital games, YouTube videos, and smart devices. Science and technology have made rapid and transformative progress in recent decades. One of these developments is the emergence of the metaverse, a rapidly expanding three-dimensional virtual space. Neal Stephenson coined the term "metaverse" in his 1992 science fiction novel Snow Crash, combining the words "meta," meaning "transcendence and virtuality," and "verse," meaning "world and universe." Enhanced by technologies such as augmented reality (AR), virtual reality (VR), and artificial intelligence, the metaverse creates a 3D virtual sphere where individuals from around the world can come together for shared social interactions. It also serves as an arena for users to participate in various social activities. In recent years, significant events such as the pandemic, conflicts, seismic activity, and climate change have led to disruptions in higher education in certain countries. Due to the pandemic, there has been a significant shift towards distance learning platforms, and students have been denied various opportunities. Distance learning is defined as "an effective form of learning that is independent of time and place. It offers individuals the ability to conveniently configure and update educational materials electronically and integrate different technologies into the learning process. These technologies can be utilized 24/7." The goal of distance education is to ensure continuity of education and increase learner satisfaction. Consequently, universities have adopted various distance learning models to address these challenges and promote their students' academic success. Using the metaverse in education is a significant application area and is widely anticipated to be very promising in the future.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student in the Department of Physiotherapy and Rehabilitation
* Having basic anatomy knowledge
* Having sufficient time and resources to participate in training and complete assessments
* Being 18 years of age or older
* Being a volunteer and providing written consent

Exclusion Criteria:

* Having previously received comprehensive palpation training
* Those at High Risk of Absence During Training
* Participants who lack the necessary hardware and internet access, especially for online and metaverse groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Instructional Materials Motivation Survey | Pre-test 1 day before intervention Post-test 1 day after intervention ends
  This scale identifies changes in students' motivation when exposed to instructional materials based on the basic components. The scale's reliability (Cronbach's alpha) internal consistency coefficient was found to be .83 for the total scale and .79 and .69 for the sub-factors, respectively. The scale's sub-dimensions are divided into attention-relevance and confidence-satisfaction. This questionnaire is self-reported and uses a five-point Likert-type scale (1 = strongly disagree, 5 = strongly agree). The potential score for the scale ranges from 24 (minimum) to 120 (maximum). Higher cumulative scores indicate increased learning motivation.
Academic Performance Assessment (exam) | 1 day after intervention ends
  Researchers will develop a 15-question multiple-choice, visual exam to assess students' proficiency in the Palpation Skills in Physiotherapy course. Before use, the test items will be administered to a separate group of students to assess validity and reliability. The test will then be administered face-to-face.

IPD SHARING:
Plan to Share IPD: No